CLINICAL TRIAL: NCT00785018
Title: In Vivo Effects of C1-esterase Inhibitor on the Innate Immune Response During Human Endotoxemia
Acronym: VECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: P. Pickkers, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: VECTOR study 2008/197
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2009-05

CONDITIONS: Endotoxemia; Inflammation; Multi Organ Dysfunction Syndrome
Keywords: Endotoxin; C1-inhibitor; Inflammation; Sepsis; Multi organ dysfunction syndrome; Complement activation
MeSH Terms: conditions — Endotoxemia; Inflammation; Angioedemas, Hereditary; Sepsis | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- C1-esterase inhibitor (Active Comparator): Endotoxin 2ng/kg followed by C1- esterase inhibitor 100 U/kg infusion
  Interventions: Drug: C1-esterase inhibitor; Drug: Endotoxin administration
- Placebo (Placebo Comparator): Endotoxin 2ng/kg followed by saline 0.9%(placebo) infusion
  Interventions: Drug: Endotoxin administration

INTERVENTIONS:
Drug: C1-esterase inhibitor — C1-esterase inhibitor 100 U/kg infusion over 30 minutes.
  Arms: C1-esterase inhibitor
Drug: Endotoxin administration — 2 ng/kg E. coli reference endotoxin 11:H 10:K negative intravenously

SUMMARY:
Excessive inflammation is associated with tissue damage caused by over-activation of the innate immune system. This can range from mild disease to extreme conditions such as multiple organ failure (MOF). In marked contrast to adaptive immunity which is very sensitive to immune modulators such as steroids, the innate immune system cannot be sufficiently targeted by currently available anti-inflammatory drugs.

We hypothesize that C1-esterase inhibitor can modulate the innate immune response.

In this study, human endotoxemia will be used as a model for inflammation. Subjects will, additionally to endotoxin, receive C1 esterase inhibitor or placebo. Blood will be sampled to determine the levels of markers of the innate immune response.

DETAILED DESCRIPTION:
Rationale:

There is an unmet need for novel therapeutic agents focused on the complications caused by acute and excessive activation of the innate immune response after injury. As this activation responds poorly to currently used therapy including inhaled steroids novel agents need to be tested, developed or applied. C1INH comprises a potential important target drug for antagonism of the excessive activation of the innate immune response during acute inflammation seen after injury. This might be achieved by inhibiting the redistribution and homing of cells to inflammatory tissues.

Before going to a clinical trial in injured human subjects we want to perform a pilot study in healthy volunteers to exploit the "human endotoxemia model". The human endotoxemia model permits elucidation of key players in this pro-inflammatory response in humans in vivo, therefore serving as a useful tool to investigate potential novel therapeutic strategies in a standardized setting. The model bears striking resemblance to LPS models in animals. These latter studies have shown that C1INH protects from neutrophil mediated disease [1-4]. Together with the finding that C1INH has been shown to be safe in the treatment of humans, we propose to use this protein in the treatment of neutrophil driven acute inflammation such as seen after injury.

Objectives:

Primary objective: The primary objective of the study is to determine the effect of C1INH on systemic activation of the innate immune response induced by LPS challenge. This response will be objectivised by measurement of enhanced TNF-α levels 90 min after LPS challenge.

Secondary Objective(s): The secondary objective of the study is to determine the effect of C1INH on redistribution of neutrophils in the human endotoxemia model.

Study design: Double-blind placebo-controlled randomized intervention study in healthy human volunteers during experimental endotoxemia.

Study population: Non-smoking healthy male volunteers, age 18-35 yrs Intervention: Subjects will receive C1INH in a dose of 100 U/kg (n=10) or placebo (n=10) 30 min after LPS administration. Pre-hydration will be performed by infusion of 1.5 L 2.5% glucose/0.45% saline solution in 1 hour before LPS administration. LPS derived from E coli O:113 will be injected (2 ng/kg iv., infusion rate 1 minute).

Main study parameters/endpoints: The main study parameter is the concentration of circulating cytokines after LPS in the absence or presence of C1INH. Secondary study parameters include the influence of C1INH on the redistribution pattern of neutrophils and neutrophil phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers (18-35 years old)

Exclusion Criteria:

* Relevant medical history
* Drug-, nicotine-, alcohol abuses
* Tendency towards fainting
* Hyper- or hypotension

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cytokines and other markers of Inflammation | 24 hrs after LPS administration
Neutrophil redistribution and phenotype | 24 hours after LPS administration
C1-inhibitor and complement concentration and activity | 24 hours after LPS administration
Hemodynamic response | 24 hours after LPS administration
Markers of Renal Injury | 24 hours after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands